CLINICAL TRIAL: NCT07127796
Title: A Non-inferiority, Randomized Double-blind Controlled Clinical Trial Comparing the Effect of Vitamin D Supplementation Derived From Fish Waste Versus Synthetic Vitamin D on Plasma Vitamin D Levels and Anthropometric and Laboratory Correlates in Healthy Subjects With Suboptimal Blood Vitamin D Levels
Brief Title: Non-inferiority RCT on Fish Waste-Derived vs. Synthetic Vitamin D Supplementation in Healthy Adults With Suboptimal Vitamin D Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Arrigo F.G. Cicero, Prof. Dr., University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-Fish Trial
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Vitamin D; Dietary Supplement
Keywords: Vitamin D; Dietary supplement; Food waist; Fish-derived vitamin D

STUDY DESIGN:
Intervention Model Description: Spontaneous interventional on dietary supplements, randomized, double-blind, parallel groups, non-inferiority, monocentric clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement - Fish-derived Vitamin D (Experimental): Fish-derived Vitamin D
  Interventions: Other: Dietary Supplement - Fish-derived Vitamin D
- Dietary supplement - Synthetic Vitamin D (Active Comparator): Synthetic Vitamin D
  Interventions: Other: Dietary Supplement - Synthetic Vitamin D

INTERVENTIONS:
Other: Dietary Supplement - Fish-derived Vitamin D — Cholecalciferol (vitamin D3). Other components: polyunsaturated fatty acids (PUFA), arabic gum, maltodextrin, pea protein hydrolisate, hard gelatine capsules.
  The fish derived vitamin D extract was obtained from sardines (Sardina pilchardus) waste ( whole fish) recovered by CNR-IRBIM (Centro Nazionale delle Ricerche-Istituto per le Risorse Biologiche e le Biotecnologie Marine) and sourced from a professional fishing fleet operating in the Adriatic Sea (Central Mediterranean). Fishes have been homogenized, freeze dried and extracted by using a Supercritical Fluid Extractor (SFE-CO2) in the laboratories of ENEA (Agenzia nazionale per le nuove tecnologie, l'energia e lo sviluppo economico sostenibile), then analyzed for the content of vitamin D3 and other bioactives by HPLC-DAD technique in the laboratories of University of Camerino and finally microencapsulated in the laboratories of University of Piemonte Orientale for the preparation of final supplement.
  Arms: Dietary supplement - Fish-derived Vitamin D
Other: Dietary Supplement - Synthetic Vitamin D — Cholecalciferol (vitamin D3). Other components: medium-chain triglycerides, alfpha-tocopherol acetate, hard gelatin capsules.
  Arms: Dietary supplement - Synthetic Vitamin D

SUMMARY:
Vitamin D is a fat-soluble vitamin with hormone-like properties, essential for numerous physiological processes in humans. It plays a central role in maintaining calcium and phosphorus homeostasis, promoting intestinal absorption of these minerals, and ensuring optimal bone mineralization. There are two main forms: vitamin D2 (ergocalciferol), primarily obtained from plant sources and supplements, and vitamin D3 (cholecalciferol), synthesized endogenously in the skin through exposure to ultraviolet B (UVB) radiation and present in animal-derived foods such as fatty fish, liver, and egg yolks. Beyond its well-known skeletal functions, vitamin D contributes to muscle contraction, immune system modulation, and regulation of cell proliferation and differentiation. Increasing evidence suggests that adequate vitamin D status may benefit cardiovascular health, glucose metabolism, and possibly reduce the risk of certain cancers, while supplementation has been associated with improved plasma lipid profiles, a relevant factor in cardiovascular risk reduction. The European Food Safety Authority has authorized various health claims for vitamin D, including its role in normal calcium and phosphorus absorption and utilization, maintenance of normal blood calcium concentrations, bone and teeth health, normal muscle function, immune defense, and reduction of the risk of falls in older adults. Despite its importance, vitamin D deficiency is recognized as a widespread public health concern across Europe, with prevalence influenced by latitude, season, skin pigmentation, and lifestyle habits. Data indicate that up to 40% of Europeans have suboptimal vitamin D levels, with deficiency rates exceeding 70% in specific high-risk groups such as elderly individuals, people with dark skin, and those with limited sun exposure. In Italy, despite abundant sunlight, vitamin D insufficiency is highly prevalent, particularly in older adults and patients with chronic illnesses. Contributing factors include urbanization, sedentary lifestyles, reduced time spent outdoors, and cultural or clothing practices limiting sun exposure. Approximately half of the Italian population is estimated to have insufficient vitamin D levels, with rates rising in the northern regions during winter months. Prolonged deficiency has severe consequences for skeletal health, including rickets in children, osteomalacia in adults, and increased risk of osteoporosis and fractures. It is also linked to a broad range of extra-skeletal effects, such as impaired immune response with greater susceptibility to infections, increased risk of chronic diseases including cardiovascular disorders, type 2 diabetes, and certain cancers, as well as muscle weakness, higher likelihood of falls, and mood disorders such as depression and seasonal affective disorder. Addressing vitamin D deficiency requires a multifaceted approach involving dietary supplementation, food fortification strategies, and public health initiatives promoting safe sunlight exposure. Severe deficiency requires pharmacological treatment with appropriately dosed medications, whereas mild deficiency can be corrected through over-the-counter supplements. In Italy, vitamin D supplements contain up to 2000 IU per day, with the recommended daily allowance for healthy adults set at 600 IU. The demand for vitamin D supplementation is reflected in market trends: the global market was valued at USD 1.69 billion in 2022 and is projected to reach USD 3.44 billion by 2031, with an estimated compound annual growth rate of 8.22% between 2023 and 2031. Against this background, the exploration of natural, sustainable sources of vitamin D, particularly from food industry by-products such as fish waste, offers an environmentally friendly alternative to synthetic forms currently dominating the market. This concept underpins the PRIN research project "Innovative and sustainable processes for the development of Vitamin D nutraceutical from fish waste: extraction, formulation and clinical study for the evaluation of its bioavailability and clinical consequence" (VITADWASTE; 2022M9JL3%; National Coordinator: Prof. Gianni Sagratini, University of Camerino), supported by the Italian Ministry of University. The project aims to develop and clinically evaluate a fish-derived vitamin D nutraceutical as a sustainable solution. Within this context, the primary objective of the present randomized, double-blind, non-inferiority clinical trial is to assess whether supplementation with fish-derived vitamin D at a dose of 600 IU per day, corresponding to 100% of the recommended daily intake for healthy adults, has an effect on plasma vitamin D levels comparable to that of an equivalent dose of standard synthetic vitamin D in healthy adults with mild vitamin D deficiency, defined by plasma concentrations between 20 and 40 ng/mL.

DETAILED DESCRIPTION:
Vitamin D is a fat-soluble vitamin with unique hormone-like properties that is indispensable for a wide range of physiological processes essential to human health and well-being. Unlike most vitamins, which must be obtained entirely from dietary sources, vitamin D can be synthesized endogenously in the skin through the action of ultraviolet B (UVB) radiation on 7-dehydrocholesterol, a process that is influenced by factors such as geographical latitude, season, time of day, skin pigmentation, age, and sunscreen use. It exists primarily in two forms: vitamin D2 (ergocalciferol), which is derived from plant-based sources and certain supplements, and vitamin D3 (cholecalciferol), which is produced in the skin and found in animal-derived foods including fatty fish, fish liver oils, egg yolks, and certain fortified products. Both forms undergo hydroxylation in the liver to 25-hydroxyvitamin D [25(OH)D], the main circulating form and clinical marker of vitamin D status, and then further hydroxylation in the kidney to form 1,25-dihydroxyvitamin D, the biologically active hormone. Vitamin D plays a central role in regulating calcium and phosphorus homeostasis by promoting intestinal absorption, maintaining optimal mineralization of the skeleton, and ensuring proper neuromuscular function. Adequate vitamin D status is necessary to prevent rickets in children, osteomalacia in adults, and to mitigate the risk of osteoporosis and fragility fractures in older populations. Beyond its skeletal effects, vitamin D exerts multiple extra-skeletal actions: it modulates innate and adaptive immune responses, influences muscle strength and coordination, regulates cell proliferation and differentiation, and has been implicated in cardiovascular function, glucose metabolism, and even cancer prevention. Recent studies have suggested that vitamin D supplementation may also improve plasma lipid profiles, thereby reducing risk factors associated with cardiovascular disease. The European Food Safety Authority (EFSA) has officially recognized and authorized several health claims for vitamin D, including its contribution to normal absorption and utilization of calcium and phosphorus, maintenance of normal blood calcium levels, preservation of normal bones, teeth, and muscle function, support for normal immune system activity, and reduction of the risk of falls in people aged 60 and over-a benefit particularly relevant for preventing fractures in the elderly. Despite these recognized benefits, vitamin D deficiency remains a major public health challenge across Europe, affecting populations regardless of climate. Overall prevalence is estimated at up to 40% in the general population, rising above 70% in high-risk groups such as elderly individuals, people with dark skin pigmentation, those who are institutionalized or housebound, and individuals with chronic illnesses or limited sun exposure. In Italy, although its Mediterranean climate might be expected to protect against hypovitaminosis D, deficiency is common, especially in northern regions during the winter months. This paradox is explained by modern lifestyle factors including urbanization, increased time spent indoors, sedentary habits, and cultural or occupational patterns that limit skin exposure to sunlight. Approximately one in two Italians has insufficient vitamin D levels, with the prevalence markedly higher in older age groups. The clinical consequences of prolonged deficiency are wide-ranging and extend well beyond skeletal fragility: children may develop rickets characterized by impaired bone growth, skeletal deformities, and muscle weakness, while adults may suffer from osteomalacia, chronic bone pain, and an increased risk of fractures due to osteoporosis. Extra-skeletal manifestations include compromised immune defense with greater susceptibility to respiratory infections, higher incidence of metabolic disorders such as type 2 diabetes, increased cardiovascular morbidity, reduced muscle strength leading to instability and falls, and mood disturbances including depression and seasonal affective disorder. Correcting vitamin D deficiency requires a combination of public health strategies including safe sun exposure campaigns, food fortification policies, and widespread access to effective supplementation. In Italy, the recommended daily allowance (RDA) for healthy adults is 600 IU, and over-the-counter supplements can contain up to 2000 IU per day for the management of mild deficiency, while severe cases require targeted pharmacological therapy at higher doses under medical supervision. The high prevalence of suboptimal vitamin D status has fueled a substantial global market for supplements, valued at USD 1.69 billion in 2022 and projected to grow to USD 3.44 billion by 2031, with a compound annual growth rate of 8.22% from 2023 to 2031. In parallel with this market expansion, there is growing interest in identifying sustainable, environmentally friendly sources of vitamin D as alternatives to the synthetic forms that dominate current production. One promising avenue is the extraction of vitamin D from food industry by-products such as fish waste, which not only offers a renewable resource but also aligns with circular economy principles and waste reduction strategies. This innovative approach is at the heart of the PRIN project "Innovative and sustainable processes for the development of Vitamin D nutraceutical from fish waste: extraction, formulation and clinical study for the evaluation of its bioavailability and clinical consequence" (VITADWASTE; 2022M9JL3%; National Coordinator: Prof. Gianni Sagratini, University of Camerino), funded by the Italian Ministry of University. The project seeks to develop a fish-derived vitamin D nutraceutical, evaluate its bioavailability in humans, and assess its clinical effects. Within this framework, the present randomized, double-blind, non-inferiority clinical trial aims to compare, in healthy subjects with mild vitamin D deficiency defined by plasma concentrations between 20 and 40 ng/mL, the effects of daily supplementation with 600 IU of fish-derived vitamin D-equivalent to 100% of the RDA for healthy adults-to those of an identical dose of standard synthetic vitamin D, with the primary endpoint being the change in plasma vitamin D levels after supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years and ≤ 60 years old
* Vitamin D plasma level between 20 and 40 ng/mL
* Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements
* Subjects agree to participate in the study and having dated and signed the informed consent form

Exclusion Criteria:

* Intake of dietary supplements or drugs containing Vitamin D
* Diagnosis of osteopenia/osteoporosis, rheumatological diseases, history of non-traumatic bone fractures
* Known diagnosis of hyperparathyroidism, hypercalcemia, severe renal failure (eGFR<30 mg/dL) Known intolerance or allergy to fish or fish derived products
* Any preventive treatments (i.e. hypocholesterolemics, antihypertensives) not stabilized in type and dose for at least 3 months
* Active pregnancy or lactation
* Any medical or surgical condition that would limit the patient adhesion to the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in plasma vitamin D concentration from baseline to 3 months after supplementation with fish-derived or synthetic vitamin D | 3 months
  The primary objective is to compare the effect of fish-based or synthetic vitamin D supplementation on the vitamin D plasma level after 3 months of treatment in healthy subjects with suboptimal vitamin D levels

SECONDARY OUTCOMES:
Change in plasma calcium concentration from baseline to 3 months after supplementation with fish-derived or synthetic vitamin D | 3 months
  Comparative evaluation of the effect of the tested dietary supplements on the calcium plasma level after 3 months of treatment in healthy subjects with suboptimal vitamin D levels
Change in plasma phosphorus concentration from baseline to 3 months after supplementation with fish-derived or synthetic vitamin D | 3 months
  Comparative evaluation of the effect of the tested dietary supplements on the phosphorus plasma level after 3 months of treatment in healthy subjects with suboptimal vitamin D levels
Change in plasma parathyroid hormone (PTH) concentration from baseline to 3 months after supplementation with fish-derived or synthetic vitamin D | 3 months
  Comparative evaluation of the effect of the tested dietary supplements on the PTH plasma level after 3 months of treatment in healthy subjects with suboptimal vitamin D levels
Change in plasma lipid profile from baseline to 3 months after supplementation with fish-derived or synthetic vitamin D | 3 months
  Comparative evaluation of the effect of the tested dietary supplements on the serum levels of plasma lipids (total cholesterol, HDL-C, LDL-C, and triglycerides) after 3 months of treatment in healthy subjects with suboptimal vitamin D levels

IPD SHARING:
Plan to Share IPD: No